CLINICAL TRIAL: NCT03996213
Title: Randomized Controlled Trial Evaluating Head-down Position Versus Leg Elevation Position Versus Supine Position During Induction of General Anesthesia and Its Effect on the Incidence of Postinduction Hypotension
Brief Title: Comparison of the Hemodynamic Effect of Three Positions During Induction of Anesthesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Hasanin, assistant professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: N-116-2018
Record Dates: First submitted 2019-06-21; First posted 2019-06-24 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Post-induction Hypotension
MeSH Terms: interventions — Head-Down Tilt

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- supine group (No Intervention): induction of anesthesia will be initiated while patient in supine position
- head down (Active Comparator): induction of anesthesia will be initiated while patient in head down position
  Interventions: Other: head down position
- leg elevation (Active Comparator): induction of anesthesia will be initiated while patient in leg elevation position
  Interventions: Other: leg elevation position

INTERVENTIONS:
Other: head down position — Head-down position will be achieved by 30 degrees tilting of the whole operating table 1-minute before induction of anesthesia. The position will be maintained for 15 minutes after induction of anesthesia
  Arms: head down
Other: leg elevation position — Leg elevation position will be achieved by raising the patient legs for 30 cm using two standard pillows positioned under the heels 1-minute before induction of anesthesia. The position will be maintained for 15 minutes after induction of anesthesia
  Arms: leg elevation

SUMMARY:
The most common methods for prevention of post-induction hypotension are preoperative fluid loading and vasopressors. Leg elevation induces an intrinsic transfusion of 150 mL blood from the lower limbs to the central fluid compartment. Leg elevation was previously reported by our group to decrease the incidence of maternal hypotension after spinal anesthesia for caesarean delivery. Passive leg raising was also reported to provide a stable hemodynamic profile during induction of anesthesia for cardiac surgery. Head-down position was previously reported as a useful measure for management of hypovolemia in various patient groups. No studies to the best of our knowledge had evaluated the compare both positions (leg elevation position and head-down position) during induction of anesthesia in non-cardiac surgery

DETAILED DESCRIPTION:
Upon arrival to the operating room, routine monitors (ECG, pulse oximetry, and non-invasive blood pressure monitor) will be applied; intravenous line will be secured, and routine pre-medications (ranitidine 50 mg and midazolam 3-5 mg) will be administrated.

Before induction of anesthesia, patients will be randomly allocated into:supine group, head-down group or leg elevation group Baseline mean arterial blood pressure will be obtained as average of 3 reading before induction of anesthesia at supine position.

Induction of anesthesia will be achieved using fentanyl (2 mcg/Kg), propofol (2 mg/Kg), and atracurium (0.5 mg/Kg). Endotracheal tube will be inserted after 3 minutes of mask ventilation. Anesthesia will be maintained by isoflurane (1-1.5%) and atracurium 10 mg increments every 20 minutes. Ringer lactate solution will be infused at a rate of 2 mL/Kg/hour.

Any episode of hypotension (defined as mean arterial pressure < 80% of the baseline reading) will be managed by 5 mcg norepinephrine. If the hypotensive episode persisted for 2 minutes, another bolus of norepinephrine will be administered.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (18-60 years), american society of anesthesiologist physical status I-II, scheduled for elective non-cardiac surgery under general anesthesia

Exclusion Criteria:

* Patients with cardiac morbidities (impaired contractility with ejection fraction < 50%, heart block, arrhythmias, tight valvular lesions), patients on antihypertensive medications, and patients with uncontrolled hypertension will be excluded from the study. Patient with decompensated respiratory disease (poor functional capacity, generalized wheezes, peripheral O2 saturation < 90% on room air), patients at increased risk of aspiration (Inadequate fasting time, chronic renal failure, diabetes mellitus, BMI≥40 kg/m2, Gastroesophageal reflux disease, Gastrointestinal obstruction, Previous upper gastrointestinal surgery and/or undergoing Upper gastrointestinal surgery), pregnant patients and patients with increased intracranial tension will be also excluded from the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 123 (Estimated)
Dates: Start 2019-07 (Estimated); Primary Completion 2019-10 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of post-induction hypotension | during 15 minutes after induction of anesthesia
  mean arterial pressure < 80% of the baseline reading

SECONDARY OUTCOMES:
Incidence of severe post-induction hypotension | during 15 minutes after induction of anesthesia
  defined as mean arterial pressure < 60% of the baseline reading
Norepinephrine consumption | during 15 minutes after induction of anesthesia
  mcg
mean arterial pressure | 1-minute intervals starting 1 minutes before induction of anesthesia till 15 minutes post-induction of anesthesia
  mmHg
heart rate | 1-minute intervals starting 1 minutes before induction of anesthesia till 15 minutes post-induction of anesthesia
  beat per minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Mohamed Hasanin, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fakhari S, Bilehjani E, Farzin H, Pourfathi H, Chalabianlou M. The effect of passive leg-raising maneuver on hemodynamic stability during anesthesia induction for adult cardiac surgery. Integr Blood Press Control. 2018 Jun 7;11:57-63. doi: 10.2147/IBPC.S126514. eCollection 2018. PMID 29922085
- [Background] Geerts BF, van den Bergh L, Stijnen T, Aarts LP, Jansen JR. Comprehensive review: is it better to use the Trendelenburg position or passive leg raising for the initial treatment of hypovolemia? J Clin Anesth. 2012 Dec;24(8):668-74. doi: 10.1016/j.jclinane.2012.06.003. PMID 23228872